CLINICAL TRIAL: NCT05529121
Title: Developing Personalized Medicine Strategies to Increase Physical Activity in Parkinson's Disease (PD) Through Digital Health Technology
Status: Completed | Type: Observational
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, James F. Morley, Co-director, Parkinson's Disease Research, Education and Clinical Center, Crescenz VAMC, Corporal Michael J. Crescenz VA Medical Center
Other Study IDs: 1616612
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Exercise; Economics, Behavioral
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Under a grant from the Department of Defense's PD program, Dr. Morley's is investigating new approaches that 1) use "gamification"- applying rules of games like point scoring, achieving silver, gold or platinum levels and competition-- to increase physical activity in PD; 2) identify whether certain PD patient respond differently to gamification interventions than others.; 3) use readily and commercially available (including Fitbits) digital health technologies to perform all study activities remotely and enable a "touchless" study where patients don't have to come in person for any studies visits. The study is underway and actively recruiting.

DETAILED DESCRIPTION:
Objectives(s): To investigate whether: 1) Protocols using gamification to increase physical activity in patients with PD employing remote intervention and assessment will be feasible and acceptable to participants; 2) Individual NMS will predict responsiveness to a gamification intervention targeting physical activity levels-facilitating a personalized approach in future efficacy studies; 3) Changes in physical activity will be associated with changes in motor symptoms, measured using the wearable Parkinson's Kinetograph (PKG)

Research Design: This is a prospective observational study. Using administrative databases and review of medical records, we will identify and remotely enroll 85 Veterans with PD on stable medication regimens into a protocol including: 1) Two week assessment of baseline activity using Fitbits; 2) a 6-week gamification intervention program targeted to a 20% increase in average daily steps; 3) 4-week follow-up period after the intervention. At baseline and following the gamification period, we will assess a variety of NMS in PD using validated questionnaires. PD motor symptoms will be assessed using the PKG (bradykinesia and motor scores) at baseline, at the end of the gamification program and after follow-up..

Methodology: All survey assessments, activity monitoring and administration of the gamification intervention will be conducted remotely using Way to Health, a web-based digital health platform developed at the University of Pennsylvania. Participants will complete surveys at the beginning of the study that quantify various sociodemographic, clinical, and geographical factors using the Way to Health platform. All participants will be mailed a Fitbit Inspire, a wearable activity tracker to be worn on the hip for 30 days to record daily steps. Participatiants will also be mailed a Parkinson's Kinetograph (PKG) to wear at baseline, at the end of the gamification program and after follow-up. Participants will sync their Fitbit data to the Way to Health platform, that has been used for previous clinical trials at the CMCVAMC. Statistical analysis: Aim 1: We will assess feasibility of the intervention using descriptive statistics; Aim 2: We will examine the association of baseline disease characteristics with response to the intervention using linear mixed effects models Aim 3: We will examine the association between changes in physical activity and motor symptoms using linear mixed effects models.

Clinical relationships: Exercise and physical activity are potential "silver bullets" in the treatment of Parkinson's disease (PD). Exercise has efficacy as a symptomatic and potentially disease-modifying therapy. However, low levels of physical activity in community-dwelling populations with PD demonstrate that exercise is not yet being used as an effective therapy. Interventions to increase activity levels of PD patients under real world conditions will have tremendous and immediate translational impact. Personalized strategies using digital health technology to increase physical activity would be highly scalable, improving the symptoms and lives of countless people living with PD The COVID19 pandemic halted most human-subjects research because of the need for face to face recruitment and visits. Traditional models of face to face recruitment and assessment are unlikely to be viable during the funding period for the proposed studies, and, perhaps, beyond. Approaches to recruitment and assessment that circumvent the need for face to face contact will have high impact.

Impact/Significance: Personalized strategies using digital health technology to increase physical activity would be highly scalable, improving the symptoms and lives of countless people living with PD.

ELIGIBILITY:
Inclusion Criteria: We will recruit Veterans within the VISN4 region who:

* Have a clinical diagnosis of PD.
* Are on a stable regimen of anti-parkinsonian medication that have not changed since the prior visit.
* Have not fallen more than once within the past year.
* To the greatest extent possible, seek to include and study Veterans with deployment, environmental, or occupational exposures as risk factors for Parkinson's disease. These will include neurotoxins (Agent Orange, Camp Lejune groundwater, Southwest Asia burn pits) and Traumatic Brain Injury, as these exposures are commonly encountered in our Veteran population and are of significant interest as risk factors for PD.

Exclusion Criteria:

* Diagnosis of an atypical parkinsonian syndrome or concomitant administration of a drug that could cause parkinsonian syndromes.
* Cardiovascular or other medical comorbidities that preclude participation in an intervention to increase physical activity
* Lack of access to a smartphone or other device (tablet or networked computer) that can be used to interface with the Fitbit app and Way to Health platform
* PD Hoehn/Yahr stage >2.5 indicating significant balance or functional impairment that would preclude participation in an intervention to increase physical activity
* Clinical diagnosis of dementia
* Active impulse control disorder

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veteran participants within the VISN4 region (a network of 9 VA medical centers and 45 outpatient clinics, covering Pennsylvania, Delaware and parts of Ohio, West Virginia, New York and New Jersey).
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility and acceptability of a "touchless" intervention to increase physical activity in patients with PD using digital health technology and behavioral economics strategies | 2026
  Protocols using gamification to increase physical activity in patients with PD employing remote intervention and assessment will be feasible and acceptable to participants. Specifically we hypothesize that subjects will: H1a) wear their activity monitor ≥ 80% of the time; H1b) successfully create a remote monitoring account and sync their device; H1c) wear and capture motor symptoms with the PKG and H1d) report high program acceptability (Intrinsic Motivation Inventory score ≥ 5)
Determine whether non-motor features predict responsiveness to a behavioral economic-based gamification intervention to increase physical activity in patients with PD | 2026
  Non-motor and features, in particular risk aversion as measured by the DOSPERT scale, will be associated with change in daily step count during the gamification intervention
Determine whether changes in physical activity in response to a gamification intervention impact PD motor symptoms measured using a remotely-monitored wearable device | 2026
  Increased activity during the gamification intervention will be associated with improvement of motor scores remotely measured using the Parkinson's Kineticgraph (PKG)

CONTACTS AND LOCATIONS:
Overall Officials: James Morley, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No